CLINICAL TRIAL: NCT05927961
Title: Spatial Proteomics Profiles of Adrenal Adenoma/Hyperplasia Leading to Primary Aldosterone
Brief Title: Spatial Proteomics Profiles of Aldosterone-producing Adenoma and Unilateral Hyperplasia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, professor, Third Military Medical University
Other Study IDs: SPP of APA/UAH
Record Dates: First submitted 2023-04-17; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Primary Aldosteronism Due to Aldosterone Producing Adenoma; Primary Aldosteronism Due to Adrenal Hyperplasia (Bilateral)
Keywords: primary aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of adrenal collected from aldosterone-producing adenoma and unilateral hyperplasia by operation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- aldosterone-producing adenoma: Histopathology shows a clear boundary between adrenal adenoma and surrounding normal tissue.
  Interventions: Diagnostic Test: histopathology
- unilateral hyperplasia: Histopathology shows no clear boundary between adrenal hyperplasia and surrounding normal tissues.
  Interventions: Diagnostic Test: histopathology

INTERVENTIONS:
Diagnostic Test: histopathology — There is a clear boundary between adrenal adenoma and surrounding normal tissue. There is no clear boundary between adrenal hyperplasia and surrounding normal tissues.

SUMMARY:
Primary aldosteronism (PA) is a common cause of secondary hypertension, which is characterized by excessive aldosterone production by the adrenal gland. Excessive aldosterone can significantly increase the risk of cardiovascular disease and stroke. Patients with aldosterone-producing adenoma (APA) or unilateral hyperplasia (UAH) can be cured by unilateral adrenalectomy. The adrenal cortex is the outer part of the adrenal gland and is subdivided into three layers- the zona glomerulosa, the zona fasciculata, and the zona reticularis. And the outermost layer is the zona glomerulosa, and it's full of cells that make the hormone aldosterone. Although it has been investigated that the main cause of APA or UAH is the mutations of different calcium ion channels, including KCNJ5, CACNA1D, CLCN2 et al, it is still unknown whether there are any other changes of other proteins in different layers. Therefore, the investigators designed the study to characterize the proteomics profiles of adrenal adenoma/hyperplasia leading to primary aldosterone and identify biomarkers for early identification of PA by using spatial proteomics. The samples from adrenal adenoma or hyperplasia will be collected and analyzed by spatial proteomics in Hangzhou Jingjie Biotechnology Co., Ltd. The differentially expressed proteins in different layers will be screened out between APA and UAH, APA and its adjacent normal tissues, and UAH and its adjacent normal tissues, respectively. And KEGG analysis will be conducted to determine enriched pathway in these differentially expressed protein, respectively.

ELIGIBILITY:
Inclusion Criteria:

* According to the 2020 guidelines for primary aldosteronism, patients with positive primary aldosteronism confirmed test;
* Patients with predominant unilateral aldosterone secretion at AVS; adrenal CT suggesting unilateral adrenal adenoma (> 0.8cm diameter) and no abnormalities in contralateral adrenal morphology.
* Patients who agreed to do the adrenalectomy.

Exclusion Criteria:

* adrenal CT suggests abnormal bilateral adrenal morphology or unilateral nodules.
* glucocorticoids can treat aldosteronism (GRA) and familial aldosteronism.
* other secondary hypertension: renal parenchymal hypertension, renal artery stenosis, Cushing syndrome, adrenal myeloid hyperplasia, aortic narrowing, obstructive sleep apnea hypoventilation syndrome.
* any other unsuitable condition for surgery.
* Patients who refused to perform adrenalectomy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We'd like to collect the samples of adrenal from primary aldosterone patients due to aldosterone-producing adenoma and unilateral hyperplasia from August 2023 to May 2024.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-25 (Estimated)

PRIMARY OUTCOMES:
Screening for the biomarkers. | After APA/UAH resection/biopsy, usually within 6 months
  Histological validation of the CYP11B2 positive area in APA and UAH by immunohistochemical staining (IHC). Some specimens will be characterized more deeply with advanced spatial proteomics technologies to identify the biomarkers.

SECONDARY OUTCOMES:
Incorporate biomarkers into the accurate and early diagnosis of PA. | 12 months
  Verifying the relationship between biomarkers and clinical presentations, including plasma aldosterone concentrations (PAC), aldosterone to rein ratio (ARR), direct renin concentration (DRC), and serum potassium, etc. Comparing the relationships between biomarkers and risk factors, including osas and family history, etc. Establishing a mathematical model for diagnosing PA through machine learning and studying the pathogenesis of PA through corresponding animal models.
Identifying the relationship between biomarkers and the prognosis of PA. | 12 months
  The alteration of blood pressure and medication status are investigated through 3 months followed up. Verifying the relationship between the biomarkers and the function of APA and UAH, as well as the prognosis of PA.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhencheng, MD, Principal Investigator — The third hospital affiliated to the Third Millitary Medical University
Locations (1):
- The Third Affiliated Hospital of the Third Military Medical University, Chongqing, China